CLINICAL TRIAL: NCT04020601
Title: The Impact of a Preoperative Nerve Block on the Consumption of Sevoflurane in Total Shoulder Arthroplasty
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00092897
Record Dates: First submitted 2019-07-10; First posted 2019-07-16 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Rotator Cuff Injuries; Anesthesia; Functional
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Ropivacaine; Glucose

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized controlled, prospective
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRE-GA (Active Comparator): 10 mL of 1% ropivacaine injection before the start of surgery and 10 ml of 5% dextrose injection at the end of surgery through the interscalene catheter
  Interventions: Drug: Ropivacaine; Drug: Dextrose
- POST-GA (Sham Comparator): 10 ml of 5% dextrose injection before the start of surgery and 1% ropivacaine injection at the end of surgery through the interscalene catheter
  Interventions: Drug: Ropivacaine; Drug: Dextrose

INTERVENTIONS:
Drug: Ropivacaine — Local anesthetic injection
Drug: Dextrose — Sham injection

SUMMARY:
Total arthroplasty surgery of the shoulder is performed under general anesthesia. Pain control for after the surgery can be achieved purely with intravenous and oral pain medication or in combination with freezing of the nerves. Nerve freezing (nerve block) placed before surgery has the potential to substantially reduce the amount of inhaled anesthetic given to the patient during surgery. This can benefit the patient by minimizing the opioid usage after surgery and also reduce cost to the system in terms of duration of hospital stay. The purpose of the study is to investigate whether the inclusion of a nerve block to the general anesthetic for total shoulder arthroplasty surgery will also reduce the amount of inhaled anesthetic and thereby lowering the environmental footprint from the anesthetic.

The investigators of the proposed study plan to quantify the amount of inhaled anesthetic used for each case and will compare how the consumption is affected by whether the nerve block is applied before or after surgery. Patients will have a nerve block catheter (interscalene catheter) placed under ultrasound-guidance prior to the induction of general anesthetic by an experienced regional anesthesiologist. The nerve block catheter will be bolused with a solution to which the anesthesiologist is blinded which will either be local anesthetic or normal saline (sham). The general anesthetic will be conducted according to a the protocol with the aim of maintaining a standard anesthetic depth monitored by patient state index (PSI). Measurements of the MAC-Value (minimum alveolar concentration) of inhaled anesthetic will be recorded every five minutes and the total amount of volatile anesthetic (in ml and ml/kg) will be noted down by a blinded observer. At the end of the case the anesthesiologist blinded to the solution will inject another solution (now a saline (sham) or local anesthetic before the patient is woken up.

DETAILED DESCRIPTION:
Following ethics approval, eligible patients meeting the inclusion/exclusion criteria will be consented in pre-assessment unit or day surgery ward at least 2 hours prior to their surgery. Patients will then be randomized into two groups:

Interscalene nerve block catheter insertion with 10 mL 1% ropivacaine injection (Treatment group) Interscalene nerve block catheter insertion with 10 mL 5% dextrose injection (Sham group)

The patient, anesthesia provider, data recorder, OR staff and Post Anaesthetic Care Unit (PACU) nurses, will be blinded at the beginning of the case. The patients consenting for the study and meeting the eligibility criteria for the study will be randomized to either group-1 (PRE-GA) or group-2 (POST-GA) . Prior to induction of general anesthesia, all patients will receive an interscalene nerve block catheter (Pajunk e-cath) inserted under ultrasound guidance using the catheter-over-needle technique by an acute pain physician who has been performing interscalene blocks under ultrasound guidance for at least 5 years. Successful catheter placement will be verified by ultrasound visualization of the injectate spread. Based on the randomization, each patient will receive a clear 10 mL syringe containing either the Treatment or the Sham solution. Patients in group PRE-GA will receive 10 ml of 1% ropivacaine through the catheter before the start of surgery and 10 ml of 5% dextrose at the end of surgery. The patients in group POST-GA will receive 10 ml of 5% dextrose before the start of surgery and 10 ml of1% ropivacaine at the end of surgery. All study medications will be prepared by the principal investigator who will be unblinded to the patient allocation. All other team members will be blinded to the group allocation.

Following the interscalene nerve block catheter insertion, all patients will receive general anesthesia with a standardized protocol using intravenous administration of fentanyl (2 mcg/kg), propofol (2 mg/kg), and rocuronium (0.6 mg/kg). General anesthesia will initially be maintained with sevoflurane at 1.0 age-adjusted Minimal Alveolar Concentration (MAC). Subsequently, the age-adjusted MAC will be titrated to achieve an intraoperative PSI target of 25-50 (Sedline, Masimo®), and intraoperative heart rate (HR) and mean blood pressure (MBP) target of +/-20% baseline values. The anaesthesiologist will have the ability to administer IV boluses of analgesic (remifentanil 0.5mcg/kg) if the Patient State Index (PSI) is >50 and/or the MBP or HR is above 20% of baseline. Vasopressors such as phenylephrine (100 mcg IV bolus) and ephedrine (5 mg IV bolus) can be used as last-line therapy to treat hypotension that is unresponsive to MAC adjustments. The age-adjusted MAC value will be recorded every 5 minutes starting at the time of skin incision until the time of skin closure. In addition, intraoperative analgesic and vasopressor usage are recorded. After the conclusion of MAC recording and prior to emergence from general anesthesia, the anaesthesiologist will be unblinded to the randomized groups, and the patients who received Sham solution will be given 10 mL of the treatment solution via the interscalene catheter to ensure patients receive adequate analgesia postoperatively.

Postoperatively, patients will be transferred to recovery area where the distribution of the sensory or motor block will then be checked and recorded 30 minutes after arriving in PACU to document the success of the block in both groups by the nurses blinded to the group allocation. The Visual Analogue Pain Scale for pain will also be recorded in PACU at 0, 15, 30 and 45 minutes. Postoperative opioid consumption, nausea and vomiting scores and pain scores over the first 24 postoperative hours will also be collected for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective shoulder arthroscopy
* Patients eligible for interscalene brachial plexus block
* All adults 18 years of age or older
* Capable to give consent

Exclusion Criteria:

* Patients who are unable to give consent
* Local anaesthetic allergy
* Hemidiaphragm paresis on the contralateral side to the block/surgery site
* Bleeding diathesis
* Coagulopathy
* Pre-existing neurological deficits
* Patients with a Body Mass Index >35
* Patients with significant comorbidities, physiological limitations, and allergies that are unable to tolerate the protocolized induction and maintenance of anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All gender identity and self-representation is eligible
Enrollment: 17 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Average age-adjusted MAC of sevoflurane | Intraoperative measurement done at the end of anesthetic
  The average age-adjusted end- tidal minimum alveolar concentration (MAC) will be calculated by averaging the end tidal MAC required to maintain the depth of anesthesia as measured by PSI between 25-50 intra-operatively. This will be compared between the two groups.

SECONDARY OUTCOMES:
Intraoperative heart rate | Intraoperative measurement
  Intraoperative heart rate (in beats/minute) will be documented at 5 minute interval and compared between the two groups
Intraoperative opioid use | Intraoperative measurement
  Intraoperative use of short acting opioid (in microgram/Kg) as per the study protocol will be recorded and compared between the two groups
Postoperative opioid use in PACU | Up to 24 postoperative hours
  Total amount of opioids (in mg of morphine equivalents) in the PACU and over the first 24 postoperative hours will be recorded and compared between the two groups
Maximum pain scores in the first 24 post-operative hours | Up to 24 postoperative hours
  Maximum pain scores will be recorded using numerical rating scale (NRS) of 0-10 (where 0=no pain and 10= maximum pain) on arrival to PACU and at 0,15,30, 45 minutes and at 24 postoperative hours and compared between the two groups
Nausea and vomiting in the first 24 post-operative hours | Up to 24 postoperative hours
  Nausea scores (on a Likert scale of 1-4 where 1 = no nausea, 2= mild nausea, 3= moderate nausea and 4= severe nausea) and incidence of vomiting will be recorded on arrival to PACU and at 0,15,30, 45 minutes and at 24 postoperative hours and will be compared between the two groups
24 hour opioid consumption | Up to 24 postoperative hours
  Frequency and total consumption of opioids (in morphine equivalents) over the first 24 postoperative hours will be recorded and compared between the two groups
The sedation score in PACU | 1st postoperative hour
  Sedation scores will be recorded at 15 minute intervals based on Ramsay sedation scale (1-6) and will be compared between the two groups
Sensory testing of nerves in the distribution of the nerve block ("Cold test") | 1st postoperative hour
  Sensory testing of the C5 and C6 dermatomes will be performed in the PACU at 30 minutes of arrival to PACU to document the success of the block
Intraoperative vasopressor usage | Intraoperative period
  Amount and frequency of the intraoperative usage of vasopressor (phenylephrine in micrograms) will be documented and compared between the two groups
Intraoperative mean blood pressure | Intraoperative period
  Intraoperative mean blood pressure (in mm Hg) will be documented at 5 minute interval and compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Vivian HY Ip, MD, Study Director — University of Alberta; Lora Pencheva, MD, Study Director — University of Alberta; Rakesh V Sondekoppam, MD, Study Chair — University of Alberta; Timur JP Özelsel, MD, DESA, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada